CLINICAL TRIAL: NCT00801346
Title: The Metabolic Syndrome in Pediatric Acute Lymphoblastic Leukemia (ALL).
Brief Title: Metabolic Syndrome in Young Patients With Acute Lymphoblastic Leukemia in Remission
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Esbenshade, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: CDR0000624471; P30CA068485 (NIH); VU-VICC-PED-0872; IRB# 081043
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Fatigue; Leukemia; Long-term Effects Secondary to Cancer Therapy in Children
Keywords: fatigue; long-term effects secondary to cancer therapy in children; childhood acute lymphoblastic leukemia in remission; B-cell childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Fatigue; Leukemia | interventions — Therapeutics

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: metabolic assessment
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: fatigue assessment and management
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about metabolic syndrome from young patients with acute lymphoblastic leukemia may help doctors learn more about the disease.

PURPOSE: This phase I trial is studying the metabolic syndrome in young patients with acute lymphoblastic leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the incidence and prevalence of the components of metabolic syndrome (e.g., obesity, hypertension, dyslipidemia, and insulin resistance) in pediatric patients with acute lymphoblastic leukemia in remission.
* To determine the trajectory of the onset of these components over a 1-year period in patients undergoing maintenance therapy.

Secondary

* To identify potential associations between components of metabolic syndrome and fatigue, health-related quality of life, family history, nutrition, and physical activity.
* To identify potential biomarkers that are associated with clinical features of metabolic syndrome.
* To evaluate whether patients will show a decrease in IGF-1 levels.

OUTLINE: This is a two-part study. Patients are enrolled in either part 1 or part 2.

* Part 1: Patients undergo physical exam measurements (e.g., body mass index, waist circumference, and blood pressure) at baseline (during maintenance course 1) and at 12 months (during maintenance course 5). Patients also undergo blood sample collection at baseline and at 12 months to measure laboratory markers (e.g., fasting lipid profile, fasting insulin and glucose, IGF-1, leptin, and adiponectin levels). Patients or their parents complete a family history questionnaire at baseline and questionnaires to assess physical activity, quality of life, nutritional intake, and fatigue at baseline and at 6 and 12 months.
* Part 2: Patients or their parents complete a family history questionnaire at baseline.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Part 1

* Diagnosis of precursor B-cell acute lymphoblastic leukemia (ALL)

  * In first remission
  * In first 3 months of maintenance therapy
* No T-cell ALL, very high-risk ALL, or infant ALL (< 1 year old at diagnosis)

Part 2

* Diagnosis of precursor B-cell or T-cell ALL

  * In first remission
* Must have been diagnosed and treated (at least to the maintenance phase) at the Division of Pediatric Oncology at the Vanderbilt-Ingram Cancer Center within the past 7 years
* No very high-risk ALL or infant ALL (< 1 year old at diagnosis)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior or concurrent cranial radiotherapy (Part 1)

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2008-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Development of components of metabolic syndrome as assessed by clinical measures (e.g., body mass index, waist circumference, and blood pressure) and laboratory measures (e.g., fasting lipid profile and fasting insulin and glucose)

SECONDARY OUTCOMES:
Diet as assessed by the Food Frequency Questionnaire at baseline and at 6 and 12 months
Family history as assessed by the Family History Questionnaire at baseline
Health-related quality of life as assessed by the Pediatric Quality of Life Inventory and the Pediatric Quality of Life Cancer Module at baseline and at 6 and 12 months
Physical activity as assessed by the Godlin Leisure Time Activity Questionnaire at baseline and at 6 and 12 months
Fatigue as assessed by the Pediatric Quality of Life Multidimensional Fatigue Survey at baseline and at 6 and 12 months
IGF-1, leptin, and adiponectin levels as assessed at baseline and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam J. Esbenshade, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee